CLINICAL TRIAL: NCT05883722
Title: Adjunctive Right Atrial Ablation for Persistent Atrial Fibrillation With Right Atrial Enlargement
Brief Title: Adjunctive Right Atrial Ablation for Persistent Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xu Liu (Other)
Collaborators: The Third Xiangya Hospital of Central South University (Other); Yangpu District Central Hospital Affiliated to Tongji University (Other)
Responsible Party: Sponsor-Investigator, Xu Liu, Prof, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KS(Y)23218
Record Dates: First submitted 2023-05-09; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation, Persistent
Keywords: catheter ablation; atrial fibrillation; Driver ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- RA group (Experimental): The RA group received adjunctive right atrial ablation in addition to left side ablation.
  Interventions: Procedure: Catheter ablation
- Control group (Active Comparator): The control group received left side ablation only.
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Procedure: Catheter ablation — The ablation approach includes: pulmonary vein isolation, left side linear ablation, left side driver ablation and right atrial driver ablation

SUMMARY:
Persistent atrial fibrillation (PerAF) can induce right atrial (RA) enlargement. Our previous study demonstrated patients with PerAF and RA enlargment may benefit from adjunctive RA ablation. Therefore, we conduct this multicenter, prospective, randomized study to confirm the value of adjunctive RA ablation.

DETAILED DESCRIPTION:
Long-term persistent atrial fibrillation (PerAF) may induce right atrial (RA) enlargement and subsequently atrial functional tricuspid regurgitation (AF-TR) at the absence of structural valvular lesion, abnormal right ventricular geometry and function. Enlarged RA and significant AF-TR may aggravate atrial remodeling and contribute to AF sustaining. Previous studies showed that RA enlargement was closely related to the recurrence of AF after catheter ablation. However, unlike the left atrium, the RA mechanism has been poorly studied and generally excluded from the therapeutic target. In an animal model of right heart disease, the RA enlargement associated with re-entrant activity serves as the prominent mechanism of AF genesis. Using sophisticated mapping techniques, recent study has confirmed that up to one-third of AF drivers are located in the right atrium. Furthermore, our previous case report also showed that the majority of patients with right atrial appendage-driven AF have concomitant RA enlargement. Therefore, it is plausible to hypothesize that the presence of RA enlargement represents the necessity of adjunctive RA ablation. Currently, the value and timing of RA intervention are still under debate. Therefore, the purpose of the present study was to testify whether patients with PerAF and RA enlargement may benefit from adjunctive RA ablation

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as persistent atrial fibrillation according to the latest clinical guidelines;
* Ineffective or intolerable to ≥1 anti-arrhythmia drug treatment.

Exclusion Criteria:

* Uncontrolled congestive heart failure;
* History of severe valve disease and/or prosthetic valve replacement;
* Myocardial infarction or stroke within 6 months;
* Severe congenital heart disease;
* EF <40%;
* Contrast agent allergy;
* The use of anticoagulant drugs is contraindicated;
* Severe lung disease;
* Left atrial thrombus confirmed by preoperative esophageal ultrasound;
* Contraindications for cardiac catheterization;
* Atrial fibrillation ablation;
* Have performed any cardiac surgery within 2 months;
* Poor general health;
* Life expectancy < 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation recurrence | 12 months
  any AF episodes lasting more than 30 seconds after the blanking period without anti-arrhythmic drugs at 12 months after a single procedure.

SECONDARY OUTCOMES:
Atrial fibrillation/atrial tachycardia recurrence | 12 months
  any documented AF/AT episode lasting more than 30 seconds after the blanking period without anti-arrhythmic drugs treatment at 12 months after a single procedure or freedom from any AF episodes lasting more than 30 seconds occurring after the blanking period without the use of anti-arrhythmic drugs at the end of study follow-up after a single procedure.